CLINICAL TRIAL: NCT01538979
Title: Phase IIb Study on the Safety and Efficacy of BM32, a Recombinant Hypoallergenic Vaccine for Immunotherapy of Grass Pollen Allergy
Brief Title: Phase II Study of Grass Pollen Allergy Vaccine BM32
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomay AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-BM32-003; 2012-000442-35 (EudraCT Number)
Record Dates: First submitted 2012-02-07; First posted 2012-02-27 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Grass Pollen Allergy
Keywords: Grass pollen allergy; Immunotherapy; Recombinant vaccine; Rhinitis, allergic, seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BM32 low dose (Experimental): 7 subcutaneous injections of 20 micrograms over two grass pollen seasons
  Interventions: Biological: BM32
- BM32 high dose (Experimental): 7 subcutaneous injections of 40 micrograms over two grass pollen seasons
  Interventions: Biological: BM32
- Placebo (Placebo Comparator): 7 subcutaneous injections over a time span of two pollen seasons
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BM32 — Subcutaneous injection of 20 micrograms of each of the protein components of BM32 adsorbed on 0.6 mg of aluminum hydroxide every 4 weeks for a total of 3 injections before each pollen season and one boost injection after pollen season
  Arms: BM32 low dose
Biological: BM32 — Subcutaneous injection of 40 micrograms of each of the protein components of BM32 adsorbed on 1.2 mg of aluminum hydroxide every 4 weeks for a total of 3 injections before each pollen season and one boost injection after pollen season
  Arms: BM32 high dose
Biological: Placebo — Subcutaneous injection of 1.2 mg of aluminum hydroxide suspension every four weeks before each pollen season and one injection after pollen season for a total of 7 injections
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy and safety of BM32 in grass pollen allergic subjects. It will test the hypothesis that either of two doses of BM32 will lead to a sustained relief off allergy symptoms over a two year study period.

DETAILED DESCRIPTION:
The present study is designed to evaluate the efficacy and safety of a treatment with the recombinant vaccine BM32 during two consecutive grass pollen seasons. Efficacy evaluation will be performed on the basis of allergy symptoms and use of relief medication as well as based on immunological parameters. After patient assessment during a screening season, patients will be randomized to one of two doses of BM32 or placebo. Patients will receive three injections of BM32 pre-season and one post-season boost injection to maintain optimal allergen specific IgG responses. Outcome will be measured after both seasons individually.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of grass pollen allergy
* Positive skin prick test reaction to grass pollen extract
* Grass pollen specific IgE and rPhl p 1/rPhl p 5 specific IgE (>3 kUA/L)
* Moderate to severe symptoms of grass pollen allergy during pollen peak

Exclusion Criteria:

* Symptomatic perennial allergies
* Atopic dermatitis
* Pregnancy or breast feeding
* Women with childbearing potential not using medically accepted birth control
* Autoimmune diseases, immune defects, immune suppression
* Immune complex induced immunopathies
* Contra indications for adrenaline
* Severe general maladies, malignancies
* Patients on long-term systematic corticosteroids, immune suppressive drugs, tranquilizers or psychoactive drugs
* Contra indication for skin prick testing
* Bronchial asthma not controlled by low dose inhaled corticosteroids
* Chronic use of beta blockers
* Participation in another clinical trial within one month prior to study
* Participation in SIT trial in 2 years prio to study
* Patients who had a previous grass pollen SIT
* Risk of non-compliance with study procedures
* Use of prohibited medications

  * Depot corticosteroids - 12 weeks prior to enrolment
  * Oral corticosteroids - 8 weeks prior to enrolment
  * High dose inhaled corticosteroids - 4 weeks prior to enrolment
  * Use of H1 antihistamines 3 days prior to enrolment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean daily combined symptom medication score (SMS)during the peak of the pollen season. | Up to 3 months
  The score will be recorded daily for the 30-45 days with the highest pollen count in each center

SECONDARY OUTCOMES:
Vital functions | Up to 22 months
Safety laboratory hematology | up to 22 months
Meal level of "well-being" measured by a visual analog scale (VAS) during grass pollen season | Up to 8 months
  The VAS will be recorded daily during the grass pollen seasons of 2013 and 2014
Number of "bad days" during the peak pollen season and the whole pollen season | Up to 8 months
  The number of bad days will be recorded daily during the grass pollen seasons of 2013 and 2014
Number of symptom-free days during the peak pollen season and the whole pollen season | Up to 8 months
  The mesure will be recorded daily during the grass pollen seasons of 2013 and 2014
Rhinoconjunctivitis quality of life evaluation by RQLQ questionnaire during pollen season | Approx. 22 months
  The questionnaire will be completed on a weekly basis during the pollen seasons of 2013 and 2014.
Mean asthma score during pollen season | Up to 8 months
  The score will be recorded on a daily basis duirng the pollen seasons of 2013 and 2014
Mean allergy specific IgG and IgE antibodies before and after vaccination | Up to 16 months
  These antibody levels will be recorded a total of five times (01/2013, 04/2013, 09/2013, 01/2014 and 04/2014)
Mean daily symptom and medication score during the whole pollen season | Up to 8 months
  The score will be recorded daily approximately during May 2013 - August 2013 and May 2014 - August 2014
Mean daily symptom score (SS) and medication score (MS) during the peak pollen season and the whole pollen season | Up to 8 months
  The scores will be recorded daily during the pollen seasons of 2013 and 2014
Skin reactivity to grass pollen extract by titrated skin prick testing | Up to 15 months
  The titrated skin prick testing will be applied a total of 4 times before and after the pollen seasons of 2013 and 2014.
Results of physical examination | up to 22 months
Safety Laboratory: Blood biochemistry | Up to 22 months
Safety laboratory: Urine analysis | up to 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ring, Prof., Study Chair — Technical University Munich, Klinik und Poliklinik für Dermatologie and Allergologie
Locations (11):
- Austria (2):
  - Medical University, Vienna, Vienna
  - Universitätsklinik für Dermatologie und Allergologie, Graz
- Allergy Network Ghent University Hospital Ghent, Dept. Otorhiolaryngologie, Ghent, Belgium
- Allergy Clinic Copenhagen University Hospital at Gentofte, Hellerup, Denmark
- Germany (5):
  - Department of Dermatology and Allergology Am Biederstein TU Munich, Munich, Bavaria
  - Allergiezentrum Charite, Berlin
  - Klinik und Poliklnik für Dermatologie und Allergologie der Universität Bonn, Bonn
  - Dept. of Dermatology and Allergology University Medical Center Gieseen and Mrbaurg GmbH, Marburg
  - Zentrum für Rhinologie/Allergologie, Wiesbaden
- Dept. of Internal Medicine Erasmus Medical Center, Rotterdam, Netherlands
- University Clinic of Respiratory and Allergic Diseases Golnik, Golnik, Slovenia